CLINICAL TRIAL: NCT07049770
Title: Efficacy of Eczeva Supplementation in Improving Skin Health
Brief Title: Eczeva Supplementation and Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zest Healthtech PLT (Industry)
Collaborators: UCSI University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEST001
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Skin; Eczema
Keywords: Eczeva; Supplements; Eczema; Natural Product; Herbal Medicine
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Intervention Model Description: This will be prospective, pre-post comparison, open-label study for a period of 20 days. FIfty subjects will be recruited in this study. The sample size calculation was based on the formula derived to determine sample size for pre-post study design (23). Total sample size needed for this study is calculated considering a type 1 error rate of 0.05, power of 80%, an expected change in standard deviation of 1.25 derived from previous study (24). The recruitment will be conducted via convenient sampling, participants will be invited via social media such as Facebook, Instagram, and WhatsApp. Participant Information Sheet (PIS) will be provided to subject, followed by consent taking before subject can access the full content of the questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental): In this arm, subjects will be required to consume Eczeva supplementation for 20 days, at the dosage of 3g once a day.
  Interventions: Dietary Supplement: Eczeva supplementation

INTERVENTIONS:
Dietary Supplement: Eczeva supplementation — Intervention contains 0.2g of eczefolia extracts, and 0.01g of rice ceramides as main active ingredients.

SUMMARY:
Eczema, also known as atopic dermatitis, is a chronic skin condition characterized by inflamed, itchy, and often dry skin. It commonly affects individuals of all ages, although it frequently begins during childhood. The causes of eczema are multifactorial, including genetic, immune, and environmental factors. Genetic mutations, such as those in the FLG gene responsible for producing filaggrin, a protein vital to skin barrier function, play a significant role (1). Immune system dysregulation, particularly an overactive response to environmental allergens, also contributes to eczema (2). Environmental triggers are diverse and include irritants like soaps, detergents, and disinfectants, as well as allergens such as pollen, pet dander, dust mites, mold, and certain foods (3-8). Climatic conditions, such as cold or dry air, and high humidity, can exacerbate symptoms, as can exposure to air pollution and chlorinated water in swimming pools (3-8). Specific skincare products containing allergens or irritants may worsen the condition. Other factors influencing eczema include infections (bacterial, viral, or fungal) (9), dietary triggers like dairy, nuts, eggs, and soy (10), and clothing choices, with materials like wool and synthetics or tight-fitting clothes aggravating symptoms through skin irritation and friction (11, 12).

Individuals with certain habits or characteristics are at a higher risk of developing eczema. A family history of eczema, asthma, or hay fever significantly increases the likelihood of the condition, as it suggests a genetic predisposition (13). Emotional stress and anxiety are known to trigger or worsen eczema symptoms (14), as are hormonal changes during pregnancy or menstruation, which can cause flare-ups (15). People who sweat excessively may experience irritation and aggravation of eczema, as the moisture can exacerbate inflammation (16). Smoking or exposure to cigarette smoke is another contributing factor, known to both trigger and worsen eczema (17). Those working in professions with frequent exposure to irritants or allergens, such as healthcare or cleaning, are at higher risk due to contact with harsh chemicals (18). Additionally, excessive hand washing can strip the skin of its natural moisture, leading to irritation and exacerbating eczema symptoms (18).

The main active ingredient in Eczeva is Melicope ptelefolia. Melicope ptelefolia, commonly known as Tenggek Burung, has been used for centuries in traditional herbal medicine to treat various skin conditions, including wounds, itches, and skin diseases (19). The plant is known for its high content of bioactive compounds, particularly 2,4,6-trihydroxy-3-geranyl acetophenone (tHGA) and 2,4,6-trihydroxy-3-prenyl acetophenone (tHPA). Among these, tHGA has shown significant potential due to its inhibitory effects on lipoxygenase (LOX) activity, suggesting its anti-inflammatory properties that may help in treating conditions like eczema (20). An in vitro study demonstrated that tHGA reduced inflammatory markers and enhanced the integrity of the skin barrier, both of which are crucial for managing inflammation-related conditions like eczema (21). Further research also indicated that tHGA could improve epithelial barrier function and reduce cell permeability in inflamed tissues, a key factor in treating eczema, which is characterized by an impaired skin barrier function (22). These findings highlight the therapeutic potential of Melicope ptelefolia in managing eczema through its anti-inflammatory and barrier-strengthening effects.

Research on the efficacy of Melicope ptelefolia supplements in improving skin health in human is remain largely unexplored. This study aims to determine the mechanism and effects of Eczeva supplements on improving the skin health among users.

ELIGIBILITY:
Inclusion Criteria:

* General healthy subject
* Aged 18 or older
* Experienced any of the following symptoms in the past 3 months:
* Skin itchiness
* Skin cracking
* Skin flaking
* Skin dryness or roughness
* Willing to comply with interventional plan
* Willing to give consent

Exclusion Criteria:

* Are pregnant or lactating
* Skin allergic due to medication, contact or seafood intakes
* Have taken dietary supplements or undergone systemic immunomodulatory or immunosuppressive therapy in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Eczema severity | Day 0 and 20
  Patient-Oriented Eczema Measure

SECONDARY OUTCOMES:
Usage of Steroids | Day 0 and 20
  Frequency and potency of the topical and oral steroids used by subject.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSI University, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years upon publication of the paper.
Access Criteria: The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request. All of the individual participant data collected during the trial, after deidentification will be shared upon reasonable request. Additional documents including study protocol, statistical analysis plan, informed consent form and clinical study report will also be made available. The data will be available immediately following publication with no end date. Data will be shared with anyone who wishes to access with reasonable request. The data can be used for any types of analyses.

REFERENCES:
- [Background] Sanioto SM, Aboulafia J. Lack of PCMB action upon the outer barrier sodium permeability in the absence of Na in toad skin. Pflugers Arch. 1985 Feb;403(2):115-9. doi: 10.1007/BF00584087. PMID 3920642